CLINICAL TRIAL: NCT01875133
Title: Effect of Altitude on Exercise Performance of Patients With Chronic Obstructive Lung Disease
Brief Title: Patients With Chronic Obstructive Pulmonary Disease At Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2013-0088
Record Dates: First submitted 2013-05-29; First posted 2013-06-11 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: airway disease; bronchitis; emphysema; lung
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: low-intermediate-high altitude (Other): Altitude exposure sequence A, 490-1630-2590m
  Interventions: Other: altitude exposure
- B: low-high-intermediate altitude (Other): Altitude exposure sequence B, 490-2590-1630 m
  Interventions: Other: altitude exposure
- C: intermediate-high-low altitude (Other): Altitude exposure sequence C, 1630-2590-490 m
  Interventions: Other: altitude exposure
- D: high-intermediate-low altitude (Other): Altitude exposure sequence D, 2590-1630-490 m
  Interventions: Other: altitude exposure

INTERVENTIONS:
Other: altitude exposure — stay at different altitudes: 490, 1630, 2590 m

SUMMARY:
The purpose of this study is to investigate the effect of a stay at moderate altitude on exercise performance of patients with chronic obstructive lung disease.

DETAILED DESCRIPTION:
Patients with moderate to severe COPD living below 800 m, will be recruited to participate in a randomized cross-over field trial evaluating the hypothesis that exercise capacity during a 4 day sojourn at moderate altitude is reduced in comparison to low altitude. Outcomes will be assessed during 2 days in Zurich (490 m, low altitude baseline), 2 days at Davos Clavadel (1650 m), and 2 days at Davos Jakobshorn (2590 m). The main outcome is the 6 minute walk distance.

ELIGIBILITY:
Inclusion Criteria:

* chronic obstructive pulmonary disease (COPD), GOLD grade 2-3
* residents at low altitude (<800 m)

Exclusion Criteria:

* Unstable condition, COPD exacerbation
* Mild (GOLD 1) or very severe COPD (GOLD 4)
* requirement for oxygen therapy at low altitude residence
* hypoventilation
* pulmonary hypertension
* more than mild or unstable cardiovascular disease
* use of drugs that affect respiratory center drive
* internal, neurologic or psychiatric disease that interfere with protocol compliance including current heavy smoking (>20 cigarettes per day), inability to perform 6 min walk test.
* previous intolerance to moderate altitude (<2600m).
* Exposure to altitudes >1500m for >2 days within the last 4 weeks before the study.
* Pregnant or nursing patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in exercise performance from baseline measured at 490 m | Change in 6 min walk distance from 490 m baseline during 2 days at 2590 m
  6 min walk distance

SECONDARY OUTCOMES:
Change in exercise performance from baseline measured at 490 m | Change in 6 min walk distance from 490 m baseline during 2 days at 1650 m
  6 min walk distance
Change in pulmonary function from baseline measured at 490 m | Change in pulmonary function from 490 m baseline during 2 days at 2590 m
  lung volumes by spirometry
Change in pulmonary function from baseline measured at 490 m | Change in pulmonary function from 490 m baseline during 2 days at 1650 m
  lung volumes by spirometry
Change in arterial blood gases from baseline measured at 490 m | Change in arterial blood gases from 490 m baseline during 2 days at 2590 m
  Arterial blood gas analysis
Change in arterial blood gases from baseline measured at 490 m | Change in arterial blood gases from 490 m baseline during 2 days at 1650 m
  Arterial blood gas analysis
Change in perceived exertion from baseline measured at 490 m | Change in perceived exertion from 490 m baseline during 2 days at 2590 m
  Borg CR10 scale at end of 6 min walk
Change in perceived exertion from baseline measured at 490 m | Change in perceived exertion from 490 m baseline during 2 days at 1650 m
  Borg CR10 scale at end of 6 min walk

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Tsogyal D Latshang, MD, Principal Investigator — University Hospital, Zürich
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Switzerland

REFERENCES:
- [Derived] Schwarz EI, Latshang TD, Furian M, Fluck D, Segitz S, Muller-Mottet S, Ulrich S, Bloch KE, Kohler M. Blood pressure response to exposure to moderate altitude in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2019 Mar 14;14:659-666. doi: 10.2147/COPD.S194426. eCollection 2019. PMID 30936690
- [Derived] Furian M, Flueck D, Latshang TD, Scheiwiller PM, Segitz SD, Mueller-Mottet S, Murer C, Steiner A, Ulrich S, Rothe T, Kohler M, Bloch KE. Exercise performance and symptoms in lowlanders with COPD ascending to moderate altitude: randomized trial. Int J Chron Obstruct Pulmon Dis. 2018 Oct 26;13:3529-3538. doi: 10.2147/COPD.S173039. eCollection 2018. PMID 30464436